CLINICAL TRIAL: NCT00712218
Title: Randomized, Multicentre Trial for Lymphadenectomy In Ovarian Neoplasms
Brief Title: Lymphadenectomy In Ovarian Neoplasms
Acronym: LION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Ursula Ghulami, KKS Marburg sponsor representative, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR OP.3
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer, FIGO stage IIB-IV
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Procedure: No Lymphadenectomy (LNE)
- B (Experimental)
  Interventions: Procedure: Lymphadenectomy (LNE)

INTERVENTIONS:
Procedure: No Lymphadenectomy (LNE) — No lymphadenectomy is performed in patients of the control group
  Arms: A
Procedure: Lymphadenectomy (LNE) — Patients allocated to the lymphadenectomy group undergo systematic lymphadenectomy in addition to surgery for complete resection. Complete mobilization of the colon by resection of the paracolic gutters is necessary for the preparation of the lymphadenectomy. Afterwards the peritoneum has to be opened until the Treitzsche's Band for visualization of the renal vein. Systematic pelvic and para-aortic lymphadenectomy is based on anatomical studies and defined according to a recently published single centre series as systematic resection of lymph nodes in the following regions [24, ].
  Arms: B

SUMMARY:
To assess the efficacy of systematic pelvic and para-aortic lymphadenectomy in patients with advanced ovarian cancer and intra-abdominal complete debulking.

Secondary: progression-free survival, complications and quality of life; Exploratory: Role of number of resected lymph nodes for primary and secondary objectives

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of invasive epithelial ovarian cancer FIGO stage IIB-IV (IV only if resectable metastasis in pleura, liver, spleen, and/or abdominal wall)
* Macroscopic complete resection
* Age: 18 - 75 years
* Patients who have given their signed and written informed consent
* Good performance status (ECOG 0/1)

Exclusion Criteria:

* Non epithelial ovarian malignancies and borderline tumors
* Intraoperative clinically suspicious lymph nodes (bulky nodes)
* Secondary invasive neoplasms in the last 5 years (except synchronal endometrial carcinoma FIGO IA G1/2, non melanoma skin cancer, breast cancer T1 N0 M0 G1/2) or with any signs of relapse or activity.
* Recurrent ovarian cancer
* Prior chemotherapy for ovarian cancer or abdominal/pelvic radiotherapy
* Diseases of the lymph system (including lymph edema of unknown origin)
* Clinical relevant dysfunctions of blood clotting (including medicamentous conditioned reasons, e.g. ASS, if not stopped at least 7 days prior to surgery)
* Any significant medical reasons, age or performance status that will not allow to perform the study procedures (estimation of investigator)
* Prior retroperitoneal lymph node dissection (systematic or sampling)
* Pregnancy
* Dementia or significantly altered mental status that would prohibit the understanding and giving of informed consent
* Any reasons interfering with regular follow-up

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2008-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival | time from randomization until death

SECONDARY OUTCOMES:
- Progression-free survival (PFS) - Quality of life (QoL) as measured by EORTC QLQ-C30, OV28 - number of resected lymph nodes | Progression-free survival time is calculated from the date of surgery until the date of first progressive disease or death, whichever occurs first or date of last contact (censored observation).

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Wagner, MD, Prof, Principal Investigator — University Marburg
Locations (59):
- Austria (4):
  - Universitaetsklinik Graz, Graz
  - Universitaetskliniken LKH Innsbruck, Innsbruck
  - AKH Wien, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- UZ Gasthuisberg, Leuven, Belgium
- Odd G1, gyn. por. klinika VFN, Prague, Czechia
- Germany (43):
  - Ostalb Klinikum Aalen, Aalen
  - Klinikum Ansbach, Ansbach
  - Hochtaunus-Kliniken gGmbH, Bad Homburg
  - SANA Klinikum Lichtenberg, Oskar-Ziehten-Krankenhaus, Berlin
  - Charite Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Malteser Krankenhaus Bonn-Rhein/Sieg, Bonn
  - Klinikum Bremen, Bremen
  - Universitaetsklinik Koeln, Cologne
  - Klinikum des Landkreises Deggendorf, Deggendorf
  - Donau-Ries Klinik Donauwoerth, Donauwörth
  - Universitaetsklinikum Carl Gustac Carus, Dresden
  - Evangelisches Krankenhaus, Düsseldorf
  - Kaiserswerther Diakonie, Florence-Nightingale Krankenhaus, Düsseldorf
  - Universitaetsklinikum Erlangen-Nuernberg, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Kliniken Essen Mitte - Evang. Huyssens Stiftung/Knappschaft GmbH, Essen
  - Klinikum der Johann-Wolfgang-Goethe Universitaet, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Fuerth, Fürth
  - Klinikum Goettingen, Göttingen
  - Klinikum der Ernst-Moritz-Arndt-Universitaet, Greifswald
  - Universitaetsklikum Hamburg-Eppendorf, Hamburg
  - Albertinen Krankenhaus, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Schleswig Holstein, Campus Kiel, Kiel
  - Asklepios Klinik, Lich
  - Klinikum Lueneburg, Lüneburg
  - Klinik für Gynäkologie, Gyn. Endokrinologie und Onkologie, Marburg
  - Klinikum der Universität Muenchen-Grosshadern, München
  - Klinikum rechts der Isar, München
  - Kliniken des Landkreises Neumarkt i. d. Opf, Klinikum Neumarkt, Neumarkt I. D. Opf
  - Klinikum Offenbach, Offenbach
  - Ortenau Klinikum St. Josefsklinik, Offenburg
  - Oberschwabenklinik Krankenhaus St. Elisabeth, Ravensburg
  - Caritas-Krankenhaus St. Josef, Regensburg
  - Frauenklinik Sana-Klinikum Remscheid GmbH, Remscheid
  - Staedtisches Klinikum Solingen, Solingen
  - Universitätsklinikum Tübingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - Dr. Horst-Schmidt-Klinik, Wiesbaden
  - Klinikum der Stadt Wolfsburg, Wolfsburg
- Italy (9):
  - Centro di Riferimento Oncologico, Aviano
  - Università Cattolica del Sacro Cuore, Campobasso
  - Ospedale di Carpi, Carpi
  - Fondazione IRCCS, Milan
  - IEO - European Institue of Oncology (Instituto Europeo di Oncologia), Milan
  - Azienda Ospedaliera S. Gerardo di Monza, Monza
  - National Cancer Institute Naples, Naples
  - Università Cattolica del Sacro Cuore, Rome
  - Ospedale Mauriziano Torino, Torino
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Harter P, Sehouli J, Lorusso D, Reuss A, Vergote I, Marth C, Kim JW, Raspagliesi F, Lampe B, Aletti G, Meier W, Cibula D, Mustea A, Mahner S, Runnebaum IB, Schmalfeldt B, Burges A, Kimmig R, Scambia G, Greggi S, Hilpert F, Hasenburg A, Hillemanns P, Giorda G, von Leffern I, Schade-Brittinger C, Wagner U, du Bois A. A Randomized Trial of Lymphadenectomy in Patients with Advanced Ovarian Neoplasms. N Engl J Med. 2019 Feb 28;380(9):822-832. doi: 10.1056/NEJMoa1808424. PMID 30811909